CLINICAL TRIAL: NCT00962260
Title: An Open-label Expanded Access Trial of Plant Cell Expressed Recombinant Human Glucocerebrosidase (prGCD) in Patients With Gaucher Disease Who Require Enzyme Replacement Therapy
Brief Title: Expanded Access Trial of Plant Expressed Recombinant Glucocerebrosidase (prGCD) in Patients With Gaucher Disease
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: PB-06-004
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Gaucher Disease
Keywords: glucocerebrosidase; enzyme replacement therapy; Gaucher disease; plant cell culture; splenomegaly; hepatomegaly; anemia; thrombocytopenia
MeSH Terms: conditions — Gaucher Disease; Splenomegaly; Hepatomegaly; Anemia; Thrombocytopenia | interventions — taliglucerase alfa

INTERVENTIONS:
Drug: Plant cell expressed recombinant glucocerebrosidase (prGCD) — Intravenous infusion every two weeks at the dose level equal to each patient's previous imiglucerase dose before reduction or discontinuation due to shortage
  Other Names: taliglucerase alfa

SUMMARY:
This is an open-label expanded access trial of prGCD in patients with Gaucher disease who require enzyme replacement therapy (ERT) and who have been treated with imiglucerase but for whom the dose has been reduced or discontinued due to shortage of the product.

DETAILED DESCRIPTION:
Gaucher disease, the most prevalent lysosomal storage disorder, is caused by mutations in the human glucocerebrosidase gene (GCD), which have been mapped to chromosome 1 q21-q31, leading to reduced activity of the lysosomal enzyme glucocerebrosidase and thereby to the accumulation of substrate glucocerebroside (GlcCer) in the cells of the monocyte-macrophage system. This accumulation leads to the visceral manifestations of hepatosplenomegaly, anemia and thrombocytopenia, as well as to the skeletal features and less frequently also to lung involvement.

prGCD is a plant cell expressed recombinant glucocerebrosidase enzyme for the treatment of Gaucher disease. Expression of proteins in plant cell culture is highly efficient, does not require post-expression modification of the protein, and is not susceptible to contamination by agents such as viruses that are pathological to humans.

prGCD safety will be observed in this treatment protocol of patients with non-neuronopathic Gaucher disease who require enzyme replacement therapy. Eligible patients will receive intravenous (IV) infusions of prGCD every two weeks. The dose of prGCD will be equal to each patient's previous imiglucerase dose before reduction or discontinuation due to shortage. The infusions will be administered at the selected medical center.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years or older
* Diagnosis of Gaucher disease treated historically with imiglucerase
* Able to provide written informed consent

Exclusion Criteria:

* Currently taking another experimental drug for any condition
* History of allergy to carrots
* Previous infusion reaction suspected to be allergic in nature to Cerezyme® or Ceredase® or receiving premedication to prevent infusion reactions
* Allergy to beta-lactam antibiotics
* Presence of any medical, emotional, behavioral or psychological condition that in the judgment of the Investigator would interfere with the patient's compliance with the requirements of the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (15):
- United States (14):
  - La Jolla Village Family Medical Group, La Jolla, California
  - University of Colorado Denver, Aurora, Colorado
  - University Research Foundation for Lysosomal Storage Diseases, Inc., Coral Springs, Florida
  - Department of Human Genetics, Emory University School of Medicine, Decatur, Georgia
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Neurogenetics, NYU at Rivergate, New York, New York
  - Division of Medical Genetics, Duke University Medical Center, Durham, North Carolina
  - Department of Medical Genetics, Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Baylor University Medical Center at Dallas, Institute of Metabolic Disease, Dallas, Texas
  - Center for Clinical Trials, Springfield, Virginia
  - University of Washington, Department of Pediatrics, Seattle, Washington
- Sha'are Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Shaaltiel Y, Bartfeld D, Hashmueli S, Baum G, Brill-Almon E, Galili G, Dym O, Boldin-Adamsky SA, Silman I, Sussman JL, Futerman AH, Aviezer D. Production of glucocerebrosidase with terminal mannose glycans for enzyme replacement therapy of Gaucher's disease using a plant cell system. Plant Biotechnol J. 2007 Sep;5(5):579-90. doi: 10.1111/j.1467-7652.2007.00263.x. Epub 2007 May 24. PMID 17524049
- [Background] Aviezer D, Brill-Almon E, Shaaltiel Y, Hashmueli S, Bartfeld D, Mizrachi S, Liberman Y, Freeman A, Zimran A, Galun E. A plant-derived recombinant human glucocerebrosidase enzyme--a preclinical and phase I investigation. PLoS One. 2009;4(3):e4792. doi: 10.1371/journal.pone.0004792. Epub 2009 Mar 11. PMID 19277123